# A Novel Cognitive Reappraisal Intervention for Suicide Prevention

IRB #1603017115

NCT03026127

ICF R33 Version 11/6/23



#### Informed Consent and HIPAA Authorization for Clinical Investigation



| Project Title: | A Novel Cognitive Reappraisal Intervention for Suicide Prevention (R33 Phase) |
|---|---|
| Research Project #: | 1603017115 |
| Principal<br>Investigator | Dimitris N. Kiosses, Ph.D |
| Arm/Group | STUDY PARTICIPANT FORM |
| Study Participant No or Number: | ame |
| , | urrently or have been (within the last 6 months) a participant in any other research<br>I Medicine, New York Presbyterian Hospital or elsewhere? If so, please inform the |
| INSTITUTION: | Weill Cornell Medicine |

### STUDY SPONSOR/FUNDING AGENCY: National Institute of Mental Health (NIMH)

#### KEY INFORMATION ABOUT THIS RESEARCH STUDY

We are asking you to choose whether to volunteer for a research study to find out if two different forms of talking therapy are effective in reducing thoughts that life is not worth living, thoughts of self-harm, thoughts of suicide, or acts of self-harm in middle aged and older adults who have been hospitalized because of a suicide attempt or thoughts of harming themselves. This page is designed to give you key information to help you decide whether to participate. We have included detailed information after this page. Ask the research team questions. If you have questions later, the contact information for the research investigator in charge of the study is below.

Purpose: What is the study about and how long will it last?

By doing this study, we hope to learn if two different forms of talking therapy are effective in reducing thoughts that life is not worth living, thoughts of self-harm, thoughts of suicide, or acts of self-harm in middle aged and older adults who have been hospitalized because of a suicide attempt or thoughts of harming themselves. Your participation in this research will last about 6 months after your discharge from the hospital.

Both study interventions are experimental, and we do not know

WEILL CORNELL MEDICAL COLLEGE CRISP, R33

IRB Protocol #1603017115 Consent version date: 10/19/2023 

#### Informed Consent and HIPAA Authorization for Clinical Investigation

| | which of these two is better. Neither study intervention is standard of care. For middle aged and older adults with depression and thoughts of self-harm, a combination of different medications and psychotherapy are considered the standards of care. |
|---|---|
| Benefits: Key reasons you might choose to volunteer | We cannot and do not guarantee that you will receive any benefits from this study. Possible benefits include the possibility that the proposed interventions will improve your mood and your thoughts that life is not worth living. We hope the information learned from this study will benefit others with depression and thoughts of self-harm in the future. For a complete description of benefits, refer to the Consent Document below. |
| Risks: Key reasons you might choose NOT to volunteer | Risks related to the therapy we are studying include: possible distress related to answering questions about your mood, thinking, and functioning, and possible fatigue or boredom as a result of repeated evaluations of your mood and mental state. You may experience a mild, temporary itching or tingling sensation in response to the electrode cap or electrode gel used when participating in the EEG that is done 4 times during the study. For a complete description of risks, refer to the Consent Document below. |
| Voluntary Participation: <b>Do you</b> have to take part in the study? | If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits or rights or access to care you would normally have if you choose not to volunteer. |
| | The person in charge of the study is Dr. Dimitris Kiosses. If you have questions, suggestions, or concerns regarding this study or you want to withdraw from the study his contact information is: 914-882-9997. If you have any questions, suggestions or concerns about your rights as a volunteer in this research, contact staff in the Weill Cornell Medicine Institutional Review Board (IRB) between the business hours of 9am and 5pm EST, Monday-Friday at 646-962-8200 or send an e-mail to <u>irb@med.cornell.edu</u> . |

This overview does not include all the information you need to know before deciding whether to take part in the study. Much additional detail is given in the full consent document, which can be found on the pages that follow. Be sure to review the rest of this consent form before deciding about participation.

WEILL CORNELL MEDICAL COLLEGE CRISP, R33

IRB Protocol #1603017115 Consent version date: 10/19/2023 

#### Informed Consent and HIPAA Authorization for Clinical Investigation

INSTITUTION: Weill Cornell Medical College

#### INTRODUCTION

You are invited to consider participating in a research study. You were selected as a possible participant in this study because you are an adult who has been hospitalized for thoughts that life is not worth living, thoughts of harming yourself, or an act of harming yourself, and depression.

Please take your time to make your decision. It is important that you read and understand several general principles that apply to all who take part in our studies:

- (a) Taking part in the study is entirely voluntary.
- (b) Personal benefit to you may or may not result from taking part in the study, but knowledge gained from your participation may benefit others;
- (c) You may decide not to participate in the study or you may decide to stop participating in the study at any time without loss of any benefits to which you are entitled.

The purpose and nature of the study, possible benefits, risks, and discomforts, other options, your rights as a participant, and other information about the study are discussed below. Any new information discovered which might affect your decision to participate or remain in the study will be provided to you while you are a participant in this study. You are urged to ask any questions you have about this study with members of the research team. You should take whatever time you need to discuss the study with your physician and family. The decision to participate or not to participate is yours. If you decide to participate, please sign and date where indicated at the end of this form.

The research study is being funded by the National Institute of Mental Health (NIMH). NIMH is providing research grant/funds for this study. Dr. Dimitris N. Kiosses is the principal investigator.

The study will take place at Weill Cornell Medicine/NewYork-Presbyterian Hospital in Westchester and in Manhattan. The study may also take place remotely, via phone or videoconference, from a location of your choosing. Weill Cornell Medicine and NewYork-Presbyterian Hospital are neither sponsors nor investigators for this study.

#### Informed Consent and HIPAA Authorization for Clinical Investigation

#### WHY IS THE STUDY BEING DONE?

The purpose of this study is to find out if two different forms of talking therapy are effective in reducing thoughts that life is not worth living, thoughts of self-harm, thoughts of suicide, or acts of self-harm in middle aged and older adults who have been hospitalized because of a suicide attempt or thoughts of harming themselves.

Psychotherapy, also known as talking therapy, is the use of psychological methods to help a person change and overcome problems in desired ways. Cognitive Reappraisal for Suicide Prevention (CRISP) differs from standard of care psychotherapy by offering a combination of emotion regulation techniques (including changing the perspective or the way you think to improve your emotional reaction). In addition to emotion regulation techniques used in the office, you will be trained to use additional strategies during times of emotional difficulties outside of the office. These strategies include the provision of environmental adaptation tools (notes, checklists, calendars, etc.), phone calls, and a tablet application called WellPATH. The tablet will be provided by the study.

Supportive Therapy incorporates standard of care approaches by using non-specific techniques to provide a supportive environment and help patients to express their feelings and focus on their strengths and abilities. These techniques include facilitating expression of affect, conveying empathy, highlighting successful experiences, and imparting optimism.

This research study is being done because effective psychotherapies are needed for middle aged and older adults who are at high risk of harming themselves, e.g., they have been hospitalized for a suicide attempt or for increased thoughts of harming themselves. Both study interventions are experimental, and we do not know which, if any, of these two is better. Neither study intervention is standard of care. For middle aged and older adults with depression and thoughts of self-harm, a combination of different medications and psychotherapy are considered the standards of care.

#### **HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?**

Participants in the study are referred to as study participants.

About 90 study participants will take part in this study; all study participants will be recruited at this site.

#### WHAT IS INVOLVED IN THE STUDY?

If you agree to participate, after you have reviewed and signed this consent form, a research assistant will conduct an assessment to find if you meet the criteria to participate. The research assistant will assess your depression, hopelessness, and thoughts of potential self-harm. If you agree and meet the study criteria, the research assistant will then conduct the rest of the interview with you for approximately 90 minutes to further assess your mood, functioning, and cognition. You will also be asked to recall situations that have triggered negative emotions in the past and link them to specific words. The assessment will also include an electroencephalogram (EEG) recording during the

WEILL CORNELL MEDICAL COLLEGE CRISP, R33

IRB Protocol #1603017115 Consent version date: 10/19/2023 

#### Informed Consent and HIPAA Authorization for Clinical Investigation

presentation of emotional and neutral words and pictures in a computer. If you feel uncomfortable, you may stop the task at any time. The EEG recording is safe and non-invasive. There are no known risks to health or safety associated with the study's EEG physiological recording procedure. There is a possibility that some participants will experience mild, temporary itching or tingling sensation in response to the electrode cap or electrode gel. However, we have well-trained personnel who will guide you and help teach you how to wash the gel from your skin after the EEG collection. Additionally, you will either have your regularly scheduled therapy session with your therapist after the EEG session, or we will schedule a debriefing session with the PI, therapist or other clinician after the EEG.

After this interview you will be "randomized" into one of two study groups: *Cognitive Reappraisal Intervention for Suicide Prevention (CRISP)* or *Supportive Therapy (ST)*. Randomization means that you are put into a group by chance, like flipping a coin. Neither you nor the researchers will choose what group you will be in, and you have an equal chance of being placed in either group.

Cognitive Reappraisal Intervention for Suicide Prevention focuses on improving the study participant's cognitive reappraisal ability, i.e. the ability to modify the appraisal of a situation in order to change its emotional significance. The goal of CRISP is to regulate negative emotion and reduce thoughts that life is not worth living or thoughts of possible self-harm. To accomplish this, the therapist will:

- 1) Teach simplified, easy to administer and use cognitive reappraisal strategies to employ in situations that trigger negative emotions.
- 2) Identify and simplify with the study participant's cognitive reappraisal techniques, rate their effectiveness on reducing negative emotions in the therapist's office, and create a plan to repeatedly employ them and assess them outside of the office. CRISP's cognitive reappraisal techniques include reappraisal of the utility of negative emotions; reappraisal of an emotionally charged trigger; "distancing" from the emotional experience and reappraisal of the emotional response to a trigger. If found helpful and participant agrees, additional environmental adaptation tools such as a tablet will be provided to the participants to help them use the distraction and other emotion regulation techniques. The tablet will be given at the beginning of the study intervention and will be returned at the end of the study intervention. The tablet may also collect data (mood ratings, duration of use, number of times the participants uses the techniques). These data will not be linked to the participant's name but to the participant's study ID. No PHI (personal health information) will be collected by the tablets.

Supportive Therapy assists study participants in expressing their feelings and focusing on their strengths and abilities in working through current difficulties. Specifically, ST employs empathic listening, reflection, emotional processing, and encouragement. The main focus of ST is:

- 1) facilitating expression of affect,
- 2) conveying to the patient that he or she is understood,
- 3) offering empathy,
- 4) highlighting success experiences, and
- 5) imparting therapeutic optimism.

ST utilizes coping skills and assets, interest in the patient, and allowance of the expression of powerful WEILL CORNELL MEDICAL COLLEGE IRB Protocol 

WEILL CORNELL MEDICAL COLLEGE CRISP, R33

#1603017115

Consent version date:

10/19/2023

#### Informed Consent and HIPAA Authorization for Clinical Investigation

emotions, facilitated by a supportive environment.

Study participants in *both* groups will receive 12 weekly sessions, after their hospital discharge, with the study therapist. Each study session will last approximately 1 hour.

Selected sessions may be audiotaped and/or videotaped for the purposes of supervision and evaluation therapist adherence to the therapy protocol, as well as for research assessment training, validity, and reliability. There will also be follow up research assessments at 6, 12, and 24 weeks (please see table below outlining activities/events in the study) after discharge. The assessments will include questions about your mood and functioning and cognition. EEG recording will be conducted at baseline, week 6, week 12, and week 24.

| | | | WEEKS (AFTER DISCHARGE) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | AT HOS | SPITAL | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 24 |
| Assessments | Admission | Discharge | | | | | | X | | | | | | X | X |
| <b>EEG Recording</b> | | Discharge | | | | | | X | | | | | | X | X |
| Therapy | | | X | X | X | X | X | X | X | X | X | X | X | X | |

Please advise the researchers of any medications you are taking. In addition, if you are taking any over- the-counter drugs or herbal supplements which you have obtained from the drug store, grocery store, etc., you should advise the researchers.

With your permission, selected sessions will be audiotaped and/or videotaped for the purposes of supervision and evaluation of therapist adherence to the therapy protocol, as well as for research assessment training, validity, and reliability. The tapes will be destroyed after the end of analyses of data. Please indicate if you do/do not wish to be audiotaped/videotaped below:

| I do wish to be audiotaped |
|---------------------------------------|
| I do <u>not</u> wish to be audiotaped |
| I do wish to be videotaped |
| I do not wish to be videotaped |

#### **HOW LONG WILL I BE IN THE STUDY?**

We think you will be in the study for approximately 6 months after your discharge from the hospital.

You can stop participating at any time. However, if you decide to stop participating in the study, we encourage you to talk to the researcher and your regular doctor first.

If you choose to not participate in the study or to leave the study, your regular care will not be affected nor will **WEILL CORNELL MEDICAL COLLEGE**IRB Protocol


WEILL CORNELL MEDICAL COLLEGE CRISP, R33

#1603017115

Consent version date:

10/19/2023

#### Informed Consent and HIPAA Authorization for Clinical Investigation

your relations with WCMC, NewYork-Presbyterian Hospital, your physicians, or other personnel. In addition, you will not lose any of the benefits to which you are entitled.

If you wish to continue to meet with the therapist or to have access to the same resources after the completion of the study, please discuss this with your therapist and Dr. Kiosses, the Principal Investigator.

Any services will be covered by you or your insurance.

#### Withdrawal by investigator, physician, or sponsor

The investigators, physicians or sponsors may stop the study or take you out of the study at any time should they judge that it is in your best interest to do so; for example, if you experience a study-related injury, if you need additional treatment or different medication, or if you do not comply with the study intervention or the study plan. They may remove you from the study for various other administrative and medical reasons. They can do this without your consent.

#### WHAT ARE THE RISKS OF THE STUDY?

Risks related to the therapy we are studying include: possible distress related to answering questions about your mood, thinking, and functioning, possible fatigue or boredom as a result of repeated evaluations of your mood and mental state, and a mild, temporary itching or tingling sensation in response to the electrode cap or electrode gel. If your condition does not improve with the study interventions that we offer in this study, you may experience increased thoughts of self-harm and may have an increased risk of self-harm and you will be referred for more intense treatment. However, you do not have to answer any questions you choose not to and you may discontinue the interview if you wish. For more information, please ask Dr. Dimitris N. Kiosses at (914) 882-9997.

#### ARE THERE ANY BENEFITS TO TAKING PART IN THE STUDY?

We cannot and do not guarantee that you will receive any benefits from this study. Possible benefits include the possibility that the proposed interventions will improve your mood and your thoughts that life is not worth living. You will also be monitored closely for depressive symptoms and thoughts of self-harm, and we will refer you for additional treatment and/or notify your physician (with your permission) if these symptoms worsen to the point where you need additional treatment. Your participation in the study will be concluded if your symptoms worsen. We hope the information learned from this study will benefit others with depression and thoughts of self-harm in the future.

#### **WHAT OTHER OPTIONS ARE THERE?**

The drug treatment that you are currently receiving will continue as is and will not be controlled by the study but by your physician. Instead of being in this study, you have the option to receive talk therapy outside this study. The study investigators will discuss additional treatment options such as drug or psychotherapy treatment that you may pursue outside of the study.

You may choose not to participate in this study.

WEILL CORNELL MEDICAL COLLEGE CRISP, R33

Rev 10-2014

IRB Protocol #1603017115 Consent version date: 10/19/2023


#### **Informed Consent and HIPAA Authorization for Clinical Investigation**

#### WHAT ABOUT CONFIDENTIALITY?

Efforts will be made to protect your medical records and other personal information to the extent allowed by law. However, we cannot guarantee absolute confidentiality. Records of study participants are stored and kept according to legal requirements and may be part of your medical record. You will not be identified personally in any reports or publications resulting from this study. Organizations that may request to inspect and/or copy your research and medical records for quality assurance and data analysis include groups such as:

- Weill Cornell Medical College and New York-Presbyterian Hospital
- The Institutional Review Board (IRB)
- The Office of Human Research Protection (OHRP)
- National Institute of Mental Health and/or their representative will have access to your files.

By signing this consent form, you authorize access to this confidential information. You also authorize the release of your medical records to Weill Cornell Medical College and NewYork-Presbyterian Hospital by any other hospitals or institutions where you might receive medical care of any kind while you are participating in this study.

If information about your participation in this study is stored in a computer, we will take the following precautions to protect it from unauthorized disclosure, tampering, or damage: computers will require a unique ID and password to prevent unauthorized disclosure, tampering, or damage of the information kept in computers. Master lists identifying patients with numbers will be kept in locked file cabinets. In addition, only personnel who are associated with the study will have access to the study specific records in the database.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### **DATA SHARING**

Data from this study may be submitted to the National Database for Clinical Trials related to Mental Illness (NDCT). NDCT is a computer system run by the National Institutes of Health that allows researchers studying mental health to collect and share information with each other. With an easier way to share, researchers hope to learn new and important things about self-harm and suicide more quickly than before.

During and after the study, the researchers will send information about your health and behavior to NDCT. However, before they send it to NDCT, they will remove information such as name, address, and phone number, and replace that information with a code number. Other researchers nationwide can then file an application with the National Institutes of Health to obtain access to your study data for research purposes. Experts at the National Institutes of Health who know how to protect health and science information will look at every request carefully to minimize risks to your privacy.

You may not benefit directly from allowing your information to be shared with NDCT. The information provided to NDCT might help researchers around the world treat patients with suicidal ideation so that they have better outcomes. NDCT will report to Congress and on its website about the different studies that researchers are conducting using NDCT data; however, NDCT will not be able to contact you individually

WEILL CORNELL MEDICAL COLLEGE CRISP, R33

IRB Protocol #1603017115 Consent version date:


10/19/2023

#### Informed Consent and HIPAA Authorization for Clinical Investigation

about specific studies. You may decide now or later that you do not want to share your information using NDCT. If so, contact the researchers who conducted this study, and they will tell NDCT, which can stop sharing the research information. However, NDCT cannot take back information that was shared before you changed your mind. If you would like more information about NDCT, this is available on-line at http://ndct.nimh.nih.gov/.

#### **CERTIFICATE OF CONFIDENTIALITY**

A Certificate of Confidentiality has been granted by the Department of Health and Human Services (DHHS). This Certificate will protect the investigators (research/study staff) from being forced to release any research data in which the study participant is identified even under a court order or subpoena. This protection is not absolute. For instance, it does not override any state requirement to report child abuse to the appropriate authorities.

## HIPAA AUTHORIZATION TO USE or DISCLOSE PROTECTED HEALTH INFORMATION FOR RESEARCH

<u>Purposes for Using or Sharing Protected Health Information:</u> If you decide to join this study, WCMC researchers need your permission to use your protected health information. If you give permission, Weill Cornell Medical College (WCMC) and/or NewYork-Presbyterian Hospital (NYPH) researchers may use your information or share (disclose) information about you for their research that is considered to be protected health information.

<u>Voluntary Choice:</u> The choice to give WCMC and/or NYPH researcher's permission to use or share your protected health information for their research is voluntary. It is completely up to you. No one can force you to give permission. However, you must give permission for WCMC and/or NYPH researchers to use or share your protected health information if you want to participate in the study. If you decline to sign this form, you cannot participate in this study, because the researchers will not be able to obtain and/or use the information they need in order to conduct their research. Refusing to give permission will not affect your ability to get usual treatment, or health care from WCMC and/or NYPH.

<u>Protected Health Information To Be Used or Shared:</u> Government rules require that researchers get your permission (authorization) to use or share your protected health information. Your medical information may be disclosed to authorized public health or government officials for public health activities when required or authorized by law. If you give permission, the researchers could use or share with the people identified in this authorization any protected health information related to this research from your medical records and from any test results which includes **demographic**, **psychological**, **physical functioning**, **and memory questionnaires**.

Other Use and Sharing of Protected Health Information: If you give permission, the researchers could also use your protected health information to develop new procedures or commercial products. They could share your protected health information with the study sponsor the WCMC Institutional Review Board, inspectors who check the research, government agencies and research study staff. The researchers could also share your protected health information with the National Institute of Mental Health.

WEILL CORNELL MEDICAL COLLEGE CRISP, R33

IRB Protocol #1603017115 Consent version date: 10/19/2023 

#### Informed Consent and HIPAA Authorization for Clinical Investigation

The information that may be shared with the sponsor and/or government agencies could include your medical record and your research record related to this study. They may not be considered covered entities under the Privacy Rule and your information would not be subject to protections under the Privacy Rule.

#### **Future Research**

You may agree to allow your data to be used for future research either within or outside WCMC and/or NYPH. If information goes to an outside entity then the privacy rule may not apply.

#### **Use of Psychotherapy Notes**

<u>What are Psychotherapy Notes for Research?</u> WCMC and/or NYPH may use or share (disclose) information about you from the doctor's notes about your psychotherapy sessions for this study that is considered to be protected health information.

#### **CANCELING AUTHORIZATION**

<u>Canceling Permission:</u> If you give the WCMC and/or NYPH researchers permission to use or share your protected health information, you have the right to cancel your permission whenever you want. However, canceling your permission will not apply to information that the researchers have already used or shared.

If you wish to cancel your permission, you may do so at any time by writing to:

Privacy Officer 1300 York Avenue, Box 303 New York, NY 10065

If you have questions about this, call: (646) 962-6930 or e-mail: privacy@med.cornell.edu

**End of Permission:** Unless you cancel it, permission for WCMC and/or NYPH researchers to use or share your protected health information for their research will never end.

#### ACCESS TO RESEARCH RECORDS

**During the course of this study, <u>vou will have access</u> to see or copy your protected health information as described in this authorization form in accordance with Weill Cornell Medical College (WCMC) and/or NewYork-Presbyterian Hospital (NYPH) policies. During your participation in this study, you will have access to your research record and any study information that is part of that record, provided that the disclosure of this information will not put your well-being in jeopardy.** 

#### WHAT ARE THE COSTS?

Study participants will not have to pay to participate in this study. You will not be responsible for any costs associated with this study. The costs of the intervention you receive during this study will be paid for by the

WEILL CORNELL MEDICAL COLLEGE CRISP, R33

IRB Protocol #1603017115

Consent version date:


10/19/2023

#### Informed Consent and HIPAA Authorization for Clinical Investigation

research project and will not be charged to you or your insurance company. No cost will be associated if you get a tablet; the tablet will be given to you for free only during the study intervention. The tablet will be returned to the PI at the end of the study intervention. You or your insurance company will be charged for continuing medical care and/or hospitalization that are not a part of the study.

#### POLICY/PROCEDURES FOR RESEARCH RELATED INJURY

The Policy and Procedure for the Sponsor are as follows: The National Institute of Mental Health will not pay for care necessitated by a research related injury.

The Policy and Procedure for Weill Cornell Medical College are as follows: We are obligated to inform you about WCMC's policy in the event injury occurs. If, as a result of your participation, you experience injury from known or unknown risks of the research procedures as described, immediate medical care and treatment.

#### POLICY/PROCEDURES FOR RESEARCH RELATED INJURY

The Policy and Procedure for the Sponsor are as follows: The National Institute of Mental Health will not pay for care necessitated by a research related injury.

The Policy and Procedure for Weill Cornell Medical College are as follows: We are obligated to inform you about WCMC's policy in the event injury occurs. If, as a result of your participation, you experience injury from known or unknown risks of the research procedures as described, immediate medical care and treatment, including hospitalization, if necessary, will be available at the usual charge for such treatment. No monetary compensation is available from WCMC or NewYork-Presbyterian Hospital. Further information can be obtained by calling the Institutional Review Board at (646) 962-8200.

#### COMPENSATION FOR PARTICIPATION

You will receive compensation for participating in this study. You will be paid \$50 for each research assessment (including EEG) at Discharge, 6, 12, and 24 weeks. In addition, you may also win up to \$10 per EEG session during one of the computer tasks. You will be paid in the form of cash, check, or gift card. You will not get paid for the screening that will determine whether you meet the study criteria. You should not expect anyone to pay you for pain, worry, lost income, or non-medical care costs that occur from taking part in this research study.

Materials or data obtained from you in this research may be used for educational or commercial purposes. It is the policy of WCMC, NewYork-Presbyterian Hospital and the National Institute of Mental Health not to provide financial compensation to you should this occur.

#### WHAT ARE MY RIGHTS AS A PARTICIPANT?

Taking part in this study is voluntary. You may choose to not take part in the study or to leave the study at any time. If you choose to not participate in the study or to leave the study, your regular care will not be affected nor

WEILL CORNELL MEDICAL COLLEGE

CRISP, R33

#1603017115 Consent version date:

10/19/2023

IRB Protocol


#### Informed Consent and HIPAA Authorization for Clinical Investigation

will your relations with the Weill Cornell Medical College, New York-Presbyterian Hospital, your physicians, or other personnel. In addition, you will not lose any of the benefits to which you are entitled.

We will tell you about new information that may affect your health, welfare, or participation in this study.

A Data Safety and Monitoring Board, an independent group of experts, will be reviewing the data from this research throughout the study. We will tell you about the new information from this or other studies that may affect your health, welfare, or willingness to stay in this study.

#### WHOM DO I CALL IF I HAVE OUESTIONS OR PROBLEMS?

For questions about the study, a research-related injury, any problems, unexpected physical or psychological discomforts, or if you think that something unusual or unexpected is happening, call Dr. Dimitris Kiosses at

914-882-9997 (cell phone), the Weill Cornell Institute of Geriatric Psychiatry at 914-997-4331, or the New York Presbyterian Hospital at 914-682-9100. Be sure to inform the physician of your participation in this study.

If you have questions about your rights as a research participant, contact the WCMC IRB Office. Direct your questions to:

Institutional Review Board at:

Address: 1300 York Avenue

Box 89

New York, New York 10065


Telephone: (646) 962-8200

IRB Protocol

#1603017115

| Project Title: A Novel Cognitive Reappra | aisal Intervention for Suicide Preven | tion (R33 Phase) |
|---|---|---|
| Principal Investigator: Dimitris N. Kioss | ees, Ph.D. | |
| RESEARCHER'S STATEMENT | | |
| I have fully explained this study to the study explained the purpose, the procedures, the bestudy. Any questions that have been raised | penefits and risks that are involved in the | his research |
| Signature of Person Obtaining the Consent (Principal Investigator or Co-investigator) | Print Name of Person | Date |
| STUDY PARTICIPANT'S STATEMEN | Γ | |
| I, the undersigned, have been informed abourisks, and I have received a copy of this consbefore I sign, and I have been told that I can participate in this study. I am free to withdradecision. This withdrawal will not in any wa and I will not lose any benefits to which I oth Dimitris Kiosses and the research staff and to unexpected or unusual symptoms. | sent. I have been given the opportunity ask other questions at any time. I volume without it is from the study at any time without it is affect my future treatment or medical nerwise am entitled. I agree to cooperate | to ask questions<br>ntarily agree to<br>need to justify my<br>all management<br>ate with Dr. |
| Signature of Study Participant | Print Name of Study Participant | Date |
| Signature of Legally Authorized Representa<br>and Relationship to participant (When A | | Date |

**Consent for Research Study**